CLINICAL TRIAL: NCT02198352
Title: A Double-blind, Placebo-controlled Single Rising Dose Tolerability Study (Parallel Groups) in Healthy Male and Female Volunteers After Intravenous Administration of BIBN 4096 BS (Dosage: 0.1 - 10 mg)
Brief Title: Study to Determine Tolerability After Intravenous Administration of BIBN 4096 BS in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1149.1
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BIBN 4096 BS - in single rising doses (Experimental)
  Interventions: Drug: BIBN 4096 BS - in single rising doses
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBN 4096 BS - in single rising doses
  Arms: BIBN 4096 BS - in single rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the present study is to obtain information about the safety, tolerability and pharmacokinetics of BIBN 4096 BS after single intravenous administration of increasing doses in healthy male and female volunteers

ELIGIBILITY:
Inclusion Criteria:

* Participants should be healthy males and females
* Age range from 21 to 50 years
* Within +- 20% of their normal weight (Broca-Index)
* All female volunteers must use a safe contraception (i.e. oral contraceptive, spiral; sterilized) and must have a negative pregnancy test
* In accordance with Good Clinical Practice (GCP) and local legislation each volunteers are supposed to give their written informed consent prior to admission to the study
* Each subject will have his medical history taken and will receive a complete medical examination (incl. blood pressure and pulse rate measurements) as well as a 12-lead Electrocardiogram (ECG) within 14 days before the first administration of the test substance.
* Haematopoietic, hepatic and renal function test will be carried out in the laboratory
* The subjects will fast for 12 hours before collection of specimens for all laboratory evaluations

Exclusion Criteria:

* Volunteers will be excluded from the study if the results of the medical examination or laboratory tests (especially those which indicate liver malfunction) are judged by the clinical investigator to differ significantly from normal clinical values
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Volunteers with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (>= 24 hours) within ten half-lives of the respective drug before enrolment in the study
* Use of any other drugs which might influence the results of the trial during the week previous to the start of the study
* Participation in another study with an investigational drug within the last two months preceding this study
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 40g/day)
* Drug abuse
* Blood donation ( >= 100 ml) within the last 4 weeks
* Excessive physical activities (e.g. competitive sports) within the last week before the study
* Pregnant and/or lactating volunteers

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 1998-06; Primary Completion 1998-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 2 months
Number of subjects with clinically significant changes in vital signs (blood pressure, pulse rate, respiratory rate) | up to 8 days after last study day
Number of subjects with abnormal changes in laboratory parameters | up to 8 days after last study day
Number of subjects with clinically relevant changes in venous-occlusion plethysmography | up to 8 hours after drug administration
Number of subjects with clinically significant changes in ECG (Electrocardiogram) | up to 8 days after last study day

SECONDARY OUTCOMES:
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours after drug administration
Cmax (Maximum measured concentration of the analyte in plasma) | up to 24 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 24 hours after drug administration
MRT (Mean residence time of the analyte in the body) | up to 24 hours after drug administration
CL (Total clearance of the analyte in plasma following extravascular administration) | up to 24 hours after drug administration
Vz (Apparent volume of distribution during the terminal elimination phase) | up to 24 hours after drug administration
Vss (Volume of distribution at steady state) | up to 24 hours after drug administration
Percentage of urinary excretion of BIBN 4096 BS | up to 24 hours after drug administration